CLINICAL TRIAL: NCT02955199
Title: Fostering Mothers' Emotionally-Responsive Parenting: A Stage III Community-Based Efficacy Trial
Brief Title: Stage III Community-based Efficacy Trial for Mothering From the Inside Out
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0407026890; 3R01DA017294 (NIH)
Record Dates: First submitted 2016-10-27; First posted 2016-11-04 (Estimated); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Addiction; Substance Abuse Drug Chronic; Child Neglect; Child Neglect Emotional; Child Abuse; Parenting; Parent-Child Problem; Parent-Child Relations; Parent / Child Problem; Parenteral Drug Abuse; Parents
MeSH Terms: conditions — Behavior, Addictive; Substance Abuse, Intravenous

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mothering From the Inside Out (Experimental): Mothering from the Inside Out (MIO) is a 12 session individual parenting therapy designed for mothers enrolled in treatment for drug and/or alcohol addiction and caring for a child between 11 and 60 months of age. MIO aims to promote their capacity for parental reflective functioning (the capacity to recognize and make sense of their own and their child's difficult emotions during challenging parenting situations).
  Interventions: Behavioral: Mothering From the Inside Out (MIO)
- Parent Education (Active Comparator): Parent Education (PE) is a 12 session individual parent counseling intervention designed for mothers enrolled in treatment for drug and/or alcohol addiction and caring for a child between 11 and 60 months of age. PE provides psycho-education about child development and parenting strategies typically available at community agencies on parenting. PE is designed to control for active treatment, treatment dose, and individualized intervention approach.
  Interventions: Behavioral: Parent Education

INTERVENTIONS:
Behavioral: Mothering From the Inside Out (MIO) — Mothering from the Inside Out (MIO) is a 12 session individual parenting therapy designed for mothers enrolled in treatment for drug and/or alcohol addiction and caring for a child between 11 and 60 months of age. MIO aims to promote their capacity for parental reflective functioning (the capacity to recognize and make sense of their own and their child's difficult emotions during challenging parenting situations).
  Other Names: Mothers and Toddlers Program; Emotionally-Responsive Parenting
  Arms: Mothering From the Inside Out
Behavioral: Parent Education — Parent Education (PE) is a 12 session individual parent counseling intervention designed for mothers enrolled in treatment for drug and/or alcohol addiction and caring for a child between 11 and 60 months of age. PE provides psycho-education about child development and parenting strategies typically available at community agencies on parenting. PE is designed to control for active treatment, treatment dose, and individualized intervention approach.
  Other Names: Mommy and Me Growing Together
  Arms: Parent Education

SUMMARY:
This is a Stage III community-based randomized clinical efficacy trial testing Mothering from the Inside Out (MIO), the first evidence-based parenting intervention designed to be delivered by addiction counselors in addiction treatment settings where parents of young children are enrolled in treatment.

DETAILED DESCRIPTION:
This is a new Stage III community-based randomized clinical efficacy trial testing Mothering from the Inside Out (MIO), the first evidence-based parenting intervention designed to be delivered by addiction counselors in addiction treatment settings where parents of young children are enrolled in treatment. MIO is a weekly individual parenting therapy developed as an enhancement to standard addiction treatment that targets the addicted mother's capacity to recognize and regulate her own emotional distress during stressful parenting situations so that she can support her child's developing capacity for emotional and behavioral regulation. This capacity, called reflective functioning (RF), is a psychological skill that promotes abstinence and also helps parents foster their young children's secure attachment. Now that MIO has demonstrated efficacy in two randomized efficacy trials, the next step will be to conduct a new Stage III community-based efficacy trial where addiction counselors are trained to deliver MIO and PE with fidelity in an addiction treatment setting and to evaluate treatment outcomes and mechanisms of change in this community setting. At the end of this trial, if MIO demonstrates efficacy, all the necessary materials will be ready to train addiction counselors across a broad range of treatment settings in a Stage IV effectiveness trial. 120 mothers in addiction treatment and caring for children ages 11 - 60 months will be randomized to 12 sessions of MIO vs PE with a trained addiction counselor and fidelity will be monitored and maintained for treatment duration. It is expected that MIO-assigned mothers will demonstrate greater improvement in the primary targeted outcome - reflective functioning at week 12 (end of treatment) and week 33 (end of follow up). It is also predicted that MIO-assigned mothers will demonstrate greater improvement in secondary outcomes, including maternal sensitivity, caregiving behavior, psychiatric distress, depression and substance use at week 12 (end of treatment) and week 33 (end of follow up). Finally, it is predicted that children of MIO-assigned mothers will demonstrate greater improvement in the secondary outcome - attachment security - at week 12 (end of treatment) and week 33 (end of follow up).

ELIGIBILITY:
Inclusion Criteria:

* English-speaking female adults (18-65 years of age)
* Receiving outpatient substance abuse treatment services at the APT Foundation
* Caring for at least one child between 11 and 60 months of age
* Express interest in receiving assistance with parenting

Exclusion Criteria:

* Actively suicidal, homicidal, or severe cognitive impairment

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2015-04; Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Maternal Reflective Functioning coded using the Parent Development Interview | Change from baseline in reflective functioning at 12 weeks
  A one hour semi-structured interview that asks mothers to describe episodes with their child that typically require the capacity for reflective functioning. The interview is coded by a rater blind to all information about the mother and her treatment assignment. The protocol is assigned a score on a scale from -1 to 9 where higher scores indicate a better capacity for reflective functioning. A score of 5 indicates average reflective functioning and a score of 3 and lower represents absence of the capacity.
Maternal Reflective Functioning coded using the Parent Development Interview | Change from baseline in reflective functioning at 33 weeks
  A one hour semi-structured interview that asks mothers to describe episodes with their child that typically require the capacity for reflective functioning. The interview is coded by a rater blind to all information about the mother and her treatment assignment. The protocol is assigned a score on a scale from -1 to 9 where higher scores indicate a better capacity for reflective functioning. A score of 5 indicates average reflective functioning and a score of 3 and lower represents absence of the capacity.

SECONDARY OUTCOMES:
Maternal Sensitivity coded with Ruth Feldman's Coding Interactive Behavior (CIB) Scales | Change from baseline in maternal sensitivity at 12 weeks
  Maternal behavior is observed during a 5 minute interaction with the target child during which they explore a set of novel toys together. Maternal Sensitivity Scale includes 12 items that are rated on a 5 point scale by a trained coder who is blind to treatment assignment and all other information about the mother-child dyad. The score range is 1 to 5 where a score of 2 and below indicates clinically significant problems and a score of 3 and higher is considered average to above average sensitivity.
Maternal Sensitivity coded with Ruth Feldman's Coding Interactive Behavior (CIB) Scales | Change from baseline in maternal sensitivity at 33 weeks
  Maternal behavior is observed during a 5 minute interaction with the target child during which they explore a set of novel toys together. Maternal Sensitivity Scale includes 12 items that are rated on a 5 point scale by a trained coder who is blind to treatment assignment and all other information about the mother-child dyad. The score range is 1 to 5 where a score of 2 and below indicates clinically significant problems and a score of 3 and higher is considered average to above average sensitivity.
Maternal Caregiving Behavior coded with the Nursing Child Assessment Satellite Training (NCAST) Teaching Scales | Change from baseline in maternal caregiving behavior at 12 weeks
  Maternal behavior is observed during a 5 minute interaction with the target child during which they explore a set of novel toys together. Maternal Sensitivity Scale includes 12 items that are rated on a 5 point scale by a trained coder who is blind to treatment assignment and all other information about the mother-child dyad. The score range is 1 to 5 where a score of 2 and below indicates clinically significant problems and a score of 3 and higher is considered average to above average sensitivity.
Maternal Caregiving Behavior coded with the Nursing Child Assessment Satellite Training (NCAST) Teaching Scales | Change from baseline in maternal caregiving behavior at 33 weeks
  Maternal behavior is observed during a 5 minute interaction with the target child during which they explore a set of novel toys together. Maternal Sensitivity Scale includes 12 items that are rated on a 5 point scale by a trained coder who is blind to treatment assignment and all other information about the mother-child dyad. The score range is 1 to 5 where a score of 2 and below indicates clinically significant problems and a score of 3 and higher is considered average to above average sensitivity.
Child Attachment coded during the Strange Situation Paradigm (SSP) | Change from baseline in child attachment status at 12 weeks
  The SSP is an experimental paradigm designed to activate attachment-based stress in the child during a series of separations and reunions with mother. The assessment takes approximately 30 minutes to complete and is rated by a trained coder who is blind to treatment assignment and all other information about the mother-child dyad (except information about known disabilities in the child). The child receives a classification of Secure, Insecure-Avoidant, Insecure-Resistant or Disorganized. The ideal classification is Secure and the most clinically significant classification is Disorganized.
Child Attachment coded during the Strange Situation Paradigm (SSP) | Change from baseline in child attachment status at 33 weeks
  The SSP is an experimental paradigm designed to activate attachment-based stress in the child during a series of separations and reunions with mother. The assessment takes approximately 30 minutes to complete and is rated by a trained coder who is blind to treatment assignment and all other information about the mother-child dyad (except information about known disabilities in the child). The child receives a classification of Secure, Insecure-Avoidant, Insecure-Resistant or Disorganized. The ideal classification is Secure and the most clinically significant classification is Disorganized.

OTHER OUTCOMES:
Addiction and Child Welfare Questionnaire (ACWQ) | Change from baseline in risk for relapse at 12 weeks
  The Addiction and Child Welfare Questionnaire is a 12 item scale that we developed to assess maternal risk for relapse. Nine items ask about recent substance use and cravings and 3 items ask about child custody status (a potential trigger for relapse). Items are rated on a binary scale and scores can range from 0 to 24 with higher scores representing higher risk for/incidence of relapse. There is no established clinical cut off for the scale.
Addiction and Child Welfare Questionnaire (ACWQ) | Change from baseline in risk for relapse at 33 weeks
  The Addiction and Child Welfare Questionnaire is a 12 item scale that we developed to assess maternal risk for relapse. Nine items ask about recent substance use and cravings and 3 items ask about child custody status (a potential trigger for relapse). Items are rated on a binary scale and scores can range from 0 to 24 with higher scores representing higher risk for/incidence of relapse. There is no established clinical cut off for the scale.
Brief Symptom Inventory | Change from baseline in psychiatric symptoms at 12 weeks
  The Brief Symptom Inventory is a well known 53-item self-report measure rated on a 4 point scale that assesses current psychiatric symptoms. Scores can range from 0 to 212. We use the T Score conversion of the Global Severity Index Composite scale to evaluate fluctuations in maternal psychiatric distress across the study. T Scores can range from 1 to 100 where a score of 60 and above indicates clinically significant psychiatric distress.
Brief Symptom Inventory | Change from baseline in psychiatric symptoms at 33 weeks
  The Brief Symptom Inventory is a well known 53-item self-report measure rated on a 4 point scale that assesses current psychiatric symptoms. Scores can range from 0 to 212. We use the T Score conversion of the Global Severity Index Composite scale to evaluate fluctuations in maternal psychiatric distress across the study. T Scores can range from 1 to 100 where a score of 60 and above indicates clinically significant psychiatric distress.
Beck Depression Inventory | Change from baseline in depression symptoms at 12 weeks
  The Beck Depression Inventory is a well known 21 item self-report measure that assesses current depressive symptoms on a 3 point Likert Scale. We use the Total Depression Score to evaluate fluctuations in maternal depression. Scores range from 0 to 63 where a score of 29 or greater indicates clinically significant depression.
Beck Depression Inventory | Change from baseline in depression symptoms at 33 weeks
  The Beck Depression Inventory is a well known 21 item self-report measure that assesses current depressive symptoms on a 3 point Likert Scale. We use the Total Depression Score to evaluate fluctuations in maternal depression. Scores range from 0 to 63 where a score of 29 or greater indicates clinically significant depression.

CONTACTS AND LOCATIONS:
Locations (1):
- The Moms 'n' Kids Program at the APT Foundation, New Haven, Connecticut, United States